CLINICAL TRIAL: NCT00363402
Title: 18FDG- PET/CT Contribution to the Assessment of Lesion Severity in Cystic Fibrosis (CF
Brief Title: 18FDG- PET/CT Contribution to the Assessment of Lesion Severity in Cystic Fibrosis (CF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, DMD, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: PETCT-HMO-CTIL
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2006-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Procedure: PET-CT

SUMMARY:
Cystic fibrosis (CF) is an autosomal recessive disorder caused by mutations in the CF trans-membrane conductance regulator (CFTR) protein. CF is the most common inherited disease of Caucasians, with a carrier frequency of 1 in 25-30 individuals. Even with the impressive advances achieved in the understanding of the molecular basis and physiopathology of CF, it remains a life-threatening disorder that causes severe lung damage and nutritional deficiencies. It is generally accepted that early therapy could delay the progression of lung disease. A number of non-invasive methods are available to monitor disease activity in CF patients; however none of the currently used tools are able to monitor real-time events. Recently high resolution computed tomography (HRCT) has been used to monitor changes in lung structure. However, HRCT does not allow differentiating between acute and chronic lesions. Positron emission tomography (PET) with 18fluoro-deoxy-glucose (FDG) has already been used in a variety of settings to visualize inflammation or infection. FDG-PET imaging appears to be a promising new tool to quantify inflammation as it can detect clinically relevant changes even when no changes or minimal ones are detected by morphologic imaging. PET/CT may consequently be used to evaluate the severity of lung inflammation/infection in CF patients, and therefore the aim of this study is to evaluate the use of PET/CT for the assessment of the severity of lung inflammation/ infection in CF patients.

DETAILED DESCRIPTION:
Cystic fibrosis patients with active lung disease will undergo a high resolution PET-CT.PET/CT scans (GE ST Discovery PET/CT scanner) will be performed 60 to 90 minutes after injection of 5 MBq/kg of FDG. PET/CT will be repeated at the end of the treatment and compared with the results of the initial scan. PET and CT will be interpreted by a certified nuclear medicine physician and by a certified radiologist, respectively, blinded to clinical data, using the PET severity score (PSS), based on the number and the intensity of FDG uptake of lung foci. Intensity of uptake will be determined by calculating the mean value for the maximum standardized uptake values (MSUV) of all foci.

(SUV = Activity concentration in ROI (region of interest) divided by injected dose / patient body weight). SUV will be measured in normal lungs to receive the normal baseline control for the calculations. The correlation with clinical data (FEV1% predicted) and sputum bacteriology will then be performed. Inflammation status will also be followed by cytokine analysis.

ELIGIBILITY:
Inclusion Criteria:CF patients with active lesions in their lungs -

Exclusion Criteria:pregnancy,

-

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Improved diagnosis of CF patients
Real-time follow up of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel